CLINICAL TRIAL: NCT00480649
Title: SUccessful Control and Clinical Effectiveness of SERETIDE Study in aSthma, a Randomised Controlled Study to Investigate the Clinical Effectiveness and Health Outcome of SERETIDE in Patients With Moderate and Severe Persistent Asthma in Korea
Brief Title: Successful Control and Clinical Effectiveness Of SERETIDE(Salmeterol/Fluticasone Propionate) Study In Asthma.(SUCCESS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 100614
Record Dates: First submitted 2007-05-30; First posted 2007-05-31 (Estimated); Last update posted 2012-11-12 (Estimated); Status verified 2012-11

CONDITIONS: Asthma
Keywords: SERETIDE; asthma; Korean; ACT
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sal/FP 50/250mcg (Active Comparator): SERETIDE 50/250
  Interventions: Drug: Salmeterol/ fluticasone propionate
- Sal/FP 50/500mcg (Active Comparator): SERETIDE 50/500
  Interventions: Drug: Salmeterol/ fluticasone propionate

INTERVENTIONS:
Drug: Salmeterol/ fluticasone propionate — 2 active arms (parellel group)
  Other Names: SERETIDE

SUMMARY:
The primary study objective is to demonstrate the clinical effectiveness of SERETIDE therapy compared to the current care in management of moderate to severe persistent asthma patients in Korea.

ELIGIBILITY:
Inclusion criteria:

* Male or female subjects aged 18 years and over who are willing to give a written consent to participate in the study.
* Subjects with a documented clinical history of reversible airways obstruction (history taking is acceptable) for at least 12 months and, in the opinion of the investigator, is able to comply with therapy and to complete the Daily Record Cards (DRCs) correctly.
* Subjects able to demonstrate the ability to effectively (physically and/or mentally) use a DISKUS (a dummy DISKUS provided for test).
* A female is eligible to enter and participate in this study
* Subjects with access to telephone (mobile or landline at home)

Exclusion criteria:

* Previous use of ICS /LABA combination inhaler (SYMBICORT (Astrazeneca) or SERETIDE) 12 weeks prior to Visit 1.
* Subjects with known or suspected hypersensitivity to inhaled steroids or Beta2-agonists.
* Subjects who have had other changes in their regular asthma medication within 2 weeks of Visit 1.
* Subjects who have had a lower respiratory tract infection within 4 weeks of Visit 1.
* Subjects who have a smoking history of 10 pack years (e.g. 10 cigarettes/day for 20 years or 20 cigarettes/day for 10 years or 40 cigarettes/day for 5 years) or more at the time of Visit 1 (Current smoker can be included even if his/her smoking history is less than 10 pack years at the time of Visit 1).
* Subjects who suffer from serious, uncontrolled diseases (including serious psychological disorders) likely to interfere with the study.
* Subjects who are on immunotherapy
* Subjects who have taken any investigational drugs within 4 weeks of Visit 1.
* Subjects who have, in the opinion of the investigator, evidence of alcohol or drug abuse.
* Females who are pregnant, lactating or are of child bearing potential and are likely to become pregnant. Females of childbearing age may be included if, in the opinion of the investigator, they are exerting adequate contraceptive precautions.
* Subjects who have previously been enrolled into this study
* Patients on regular oral or parenteral steroid therapy in the last 4 weeks or more than 3 courses of steroid in the last 6 months
* Subjects who have FEV1 or PEFR of less than 50% predictive value.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2004-01; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint for this trial is mean morning PEFR LOCF at 52 weeks as collected in diary cards over the last 2 weeks preceding the 52 weeks visit. | 52 weeks after randomization

SECONDARY OUTCOMES:
Secondary measures of efficacy consist of clinical efficacy and health outcome measurements. | 52 weeks after randomization

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (8):
- South Korea (8):
  - GSK Investigational Site, Anyang-si
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Jeonju
  - GSK Investigational Site, Junjoo-Si
  - GSK Investigational Site, Kyungki-Do Anyang-si
  - GSK Investigational Site, Kyungki-Do
  - GSK Investigational Site, Pusan
  - GSK Investigational Site, Seoul

REFERENCES:
- [Background] Jung KS, Uh ST, Lee YC, Shim JJ, Park SK, Williams AE, Chan R. Comparison of the clinical efficacy and safety of salmeterol/fluticasone propionate versus current care in the management of persistent asthma in Korea. Curr Med Res Opin. 2008 Dec;24(12):3571-82. doi: 10.1185/03007990802588737. PMID 19032138